CLINICAL TRIAL: NCT06377332
Title: Biomarkers of Dementia in Chronic Sleep and Breathing Disorders
Acronym: ORACLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Sponsor
Other Study IDs: X23-0330
Record Dates: First submitted 2023-11-06; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: COPD; Overlap Syndrome; OSA
Keywords: Biomarkers; Observational; Cross-Sectional
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Magnetic Resonance Imaging; Blood Specimen Collection; Surveys and Questionnaires; Respiratory Function Tests; Mental Status and Dementia Tests; Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood collection and analyses will involve apolipoprotein 4 (APOE4) with consent
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Chronic Obstructive Pulmonary Disease (COPD): Males and females; Aged 40-65 years; COPD confirmed by diagnosis or a positive lung function test (GOLD 2 minimum, FEV1
  ≥50%, < 80% predicted; FEV1/FVC < 0.7); 10-pack year smoking history; Able to perform neuropsychological and cognitive testing; Fluent in English.
  Interventions: Diagnostic Test: High density electroencephalogram (HdEEG); Diagnostic Test: Functional near infrared spectroscopy (fNIRS); Diagnostic Test: Magnetic resonance imaging (MRI); Biological: Blood collection; Diagnostic Test: Neuropsychological battery; Other: Questionnaires; Diagnostic Test: Pulmonary Function Test (PFT); Other: Cognitive Assessment; Diagnostic Test: Polysomnogram (PSG)
- Overlap Syndrome (OVS): Males and females; Aged 40-65 years; Oximetry confirmed moderate to severe OSA based on the oxygen desaturation index (ODI) ≥15/hr OR defined by polysomnography (PSG) AHI of ≥ 15 COPD confirmed by diagnosis or a positive lung function test (GOLD 2 minimum, FEV1
  ≥50%, < 80% predicted; FEV1/FVC < 0.7); 10-pack year smoking history; Able to perform neuropsychological and cognitive testing; Fluent in English.
  Interventions: Diagnostic Test: High density electroencephalogram (HdEEG); Diagnostic Test: Functional near infrared spectroscopy (fNIRS); Diagnostic Test: Magnetic resonance imaging (MRI); Biological: Blood collection; Diagnostic Test: Neuropsychological battery; Other: Questionnaires; Diagnostic Test: Pulmonary Function Test (PFT); Other: Cognitive Assessment; Diagnostic Test: Polysomnogram (PSG)
- Obstructive Sleep Apnoea (OSA): Males and females; Aged 40-65 years; Oximetry confirmed moderate to severe OSA based on the oxygen desaturation index (ODI) ≥15/hr OR defined by polysomnography (PSG) AHI of ≥ 15. Able to give informed consent; Ability to perform neuropsychological and cognitive testing; Fluent in English.
  Interventions: Diagnostic Test: High density electroencephalogram (HdEEG); Diagnostic Test: Functional near infrared spectroscopy (fNIRS); Diagnostic Test: Magnetic resonance imaging (MRI); Biological: Blood collection; Diagnostic Test: Neuropsychological battery; Other: Questionnaires; Diagnostic Test: Pulmonary Function Test (PFT); Other: Cognitive Assessment; Diagnostic Test: Polysomnogram (PSG)
- Control: Males and females; Aged 40-65 years; Able to give informed consent; Able to perform neuropsychological and cognitive testing; Fluent in English.
  Interventions: Diagnostic Test: High density electroencephalogram (HdEEG); Diagnostic Test: Functional near infrared spectroscopy (fNIRS); Diagnostic Test: Magnetic resonance imaging (MRI); Biological: Blood collection; Diagnostic Test: Neuropsychological battery; Other: Questionnaires; Diagnostic Test: Pulmonary Function Test (PFT); Other: Cognitive Assessment; Diagnostic Test: Polysomnogram (PSG)

INTERVENTIONS:
Diagnostic Test: High density electroencephalogram (HdEEG) — High-density electroencephalography (HdEEG) will be utilised in the investigation of sleep-mediated neuronal functions in controls, OSA, COPD and overlap syndrome and the association with accelerated brain ageing and cognitive impairment.
Diagnostic Test: Functional near infrared spectroscopy (fNIRS) — Functional near infrared spectroscopy (fNIRS) is one of the most advanced techniques in measuring brain oxygen content and hemodynamic activity. This information indirectly displays neuronal activity and provides a novel opportunity understand brain oxygenation, neurodegenerative diseases, and cognitive function.
Diagnostic Test: Magnetic resonance imaging (MRI) — Magnetic resonance imaging (MRI) will be utilised to assess potential structural neuronal changes associated with neurodegenerative disease in those with COPD, OSA and overlap syndrome. MRI has the capacity to provide vital information regarding neuroimaging standards in cerebral vascular damage such as white matter hyperintensities (WMH), lacunes, cerebral microbleeds, brain atrophy and subcortical infarct. Through the utility of MRI sequences such as T1 and T2 weighted imaging, diffusion weighted imaging (DWI) and fluid-attenuated inversion recovery (FLAIR) and resting-state fMRI (rs-fMRI), the investigators will assess neurodegenerative-related structural brain changes in individuals with COPD, OSA and overlap syndrome and examine the differences between these target groups.
Biological: Blood collection — A fasting 50mL blood sample will be collected at the experimental visit in the morning following the overnight sleep study. Blood samples will be processed after collection and stored at -80 degrees for future batch analyses. Analyses will include markers for inflammation and dementia including but not limited to ptau217 and beta amyloid. Routine blood analyses will be conducted on 17.5mL of the sample collected for baseline measures. Routine blood analyses includes lipid profile, glucose studies, insulin, high-sensitivity C-reactive protein (hs-CRP), iron studies, thyroid function, b12/folate, homocysteine, prolactin, calcium, full blood count and biochemistry panel for the OSA, COPD and overlap syndrome groups.
  Routine blood analyses for controls include glucose studies, lipid profile, hs-CRP and biochemistry panel.
Diagnostic Test: Neuropsychological battery — A. Montreal Cognitive Assessment (MoCA):
  B. Test of Premorbid Functioning (TOPF):
  C. Rey Auditory Verbal Learning Test (RAVLT):
  D. D-KEFS Colour Word Interference Test (D-CWIT):
  E. Trail Making Test (TMT):
  F. Symbol Digit Modalities Test (SDMT) - Oral Version:
  G. RAVLT 20-minute recall
  H. Controlled Oral Word Association Test (COWAT):
Other: Questionnaires — 1. Epworth Sleepiness Scale (ESS)
  2. PROMIS sleep questionnaire 8a,
  3. PROMIS sleep questionnaire 8b
  4. EQ-5D-5L
  5. Insomnia Severity Index (ISI)
  6. Pittsburgh Sleep Quality Index (PSQ-I)
  7. St George's Respiratory Questionnaire (SGRQ)
  8. COPD Assessment Test (CAT)
Diagnostic Test: Pulmonary Function Test (PFT) — Full pulmonary function testing will be conducted in control, COPD, OSA and overlap syndrome groups. Full lung function testing will include spirometry with pre and post bronchodilator, oscillometry, lung diffusion testing (DLCO) and lung volumes.
Other: Cognitive Assessment — The following cognitive assessments will be administered using a digital format on CANTAB:
  1. Motor Screening Task (MOT) Used to assess sensorimotor function and comprehension and is applicable in the assessment of general cognitive function, Alzheimer's disease and cerebrovascular disease. This task acts as a practice trial for the subsequent tasks.
  2. Reaction Time (RTI) Used to assess processing and psychomotor speed and is applicable in the assessment of general cognitive function and Alzheimer's disease.
  3. Paired Associate Learning (PAL) Used to assess visual episodic memory and is applicable in the assessment of general cognitive function, Alzheimer's disease, Parkinson's disease and cerebrovascular disease.
  4. Spatial Working Memory (SWM) Used to assess working memory and strategy and is applicable in the assessment of general cognitive function, Alzheimer's disease and cerebrovascular disease.
Diagnostic Test: Polysomnogram (PSG) — During the sleep study, physiological signals are recorded to capture eye movements (electrooculogram, EOG) and chin muscle movements (electromyogram, EMG). A nasal airflow piece, two respiratory inductance plethysmography (RIP) bands and an oximeter probe on the finger will monitor breathing and oxygen levels in the blood. Electrocardiogram (ECG), leg movements, sleeping position and snoring are also recorded.

SUMMARY:
Chronic obstructive pulmonary disease (COPD), obstructive sleep apnoea (OSA) and overlap syndrome are associated with obstructions in breathing and disturbed sleep.

Chronic breathing disruptions and poor sleep may lead to cognitive impairment and brain changes linked with early neurodegenerative processes. As such, identifying early markers of cognitive impairment and dementia risk in individuals with chronic respiratory and sleep breathing disorders is crucial for understanding how these diseases may contribute to accelerated brain ageing. This study will comprehensively measure sleep, lung function, cognitive performance and blood-based markers of dementia risk and inflammation. The investigators will use innovative technologies to identify biomarkers of cognitive impairment and dementia risk in people with chronic sleep and breathing disorders. The investigators will also investigate the relationships between disrupted sleep and abnormal breathing and the brain. This research may also inform future early interventions to improve cognition and brain health in chronic sleep and respiratory disease.

DETAILED DESCRIPTION:
Neurodegeneration that is present in dementia is caused, in part, by neuroinflammation, cerebral vascular damage and oxidative stress. Intermittent hypoxia and hypercapnia, as seen in patients with chronic obstructive pulmonary disease (COPD), obstructive sleep apnoea (OSA) and overlap syndrome, cause neuroinflammation and sleep fragmentation. As a result, key biomarkers of cytokine tumour necrosis factor-alpha (TNF-a), C-reactive protein (CRP), eosinophils, CD8+ and CD4+ T cells, interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-1 beta (IL-1B), nuclear factor kappa beta (NF-kB) and hypoxia-inducible factor (HIF) infiltrate the central nervous system (CNS), perpetuating neuroinflammation through the presence of microglia which cause oxidative and nitrosative stress.

Key inflammatory and dementia-based biomarkers will be collected in the investigation of this association including but not limited to Aβ40/42 ratio and ptau217.

This study consists of an observational cross-sectional design with the utilisation of blood collection, lung function testing, MRI, HdEEG, fNIRS and neurocognitive assessment. Participants will be selected into the study differentially based on the target group, with OSA criteria requiring an ODI > 15, COPD criteria requiring a GOLD 2 minimum, FEV1 ≥50%, < 80% predicted; FEV1/FVC < 0.7 with a 10- pack year smoking history and overlap syndrome criteria requiring a combination of ODI > 15 and GOLD 2 minimum, FEV1 ≥50%, < 80% predicted; FEV1/FVC < 0.7, with a 10-pack year smoking history. Participants will be 40 to 65 years old. Controls will have no diagnosis of OSA, COPD or overlap syndrome and have an English fluency. In order to test the hypotheses, the design of a cross-sectional study will allow us to a) examine the relationships between sleep and breathing metrics and cognition and blood-based markers of dementia pathology b) examine the relationships between potential intermediates of compromised sleep and breathing with the primary cognitive and dementia risk outcomes c) compare sleep, lung function, brain health, cognition and inflammatory markers between OSA, COPD, overlap syndrome and control groups.

ELIGIBILITY:
Inclusion Criteria:

Control:

1. Males and females;
2. Aged 40-65 years;
3. Able to give informed consent;
4. Able to perform neuropsychological and cognitive testing;
5. Fluent in English.

OSA:

1. Males and females;
2. Aged 40-65 years;
3. Oximetry confirmed moderate to severe OSA based on the oxygen desaturation index (ODI) ≥15/hr;
4. Able to give informed consent;
5. Ability to perform neuropsychological and cognitive testing;
6. Fluent in English.

COPD:

1. Males and females;
2. Aged 40-65 years;
3. COPD confirmed by diagnosis or a positive lung function test (GOLD 2 minimum, FEV1

   ≥50%, < 80% predicted; FEV1/FVC < 0.7);
4. 10-pack year smoking history;
5. Able to perform neuropsychological and cognitive testing;
6. Fluent in English.

Overlap Syndrome:

1. Males and females;
2. Aged 40-65 years;
3. Oximetry confirmed moderate to severe OSA based on the oxygen desaturation index (ODI) ≥15/hr;
4. COPD confirmed by diagnosis or a positive lung function test (GOLD 2 minimum, FEV1

   ≥50%, < 80% predicted; FEV1/FVC < 0.7);
5. 10-pack year smoking history;
6. Able to perform neuropsychological and cognitive testing;
7. Fluent in English.

Exclusion Criteria:

1. Dementia diagnosis;
2. At home or overnight oxygen therapy;
3. Asthma diagnosis (identified with lung function bronchodilator);
4. Current antipsychotic use;
5. BMI > 40;
6. PAP use or OSA treatment in the last 2 months;
7. Recent COPD exacerbation with change in symptomology (hospitalisation and/or steroids and/or antibiotics) within 6 weeks;
8. Awake supine oxygen saturations of < 93%;
9. Sleep disorders including narcolepsy, idiopathic hypersomnia (IH), moderate-severe restless leg syndrome (RLS) or REM behaviour disorder (RBD);
10. Other major comorbidities (other lung diseases, neurodegenerative disease, brain injury, severe mental illness, PTSD);
11. Uncontrolled depression (impacting daily life, no use of medications or engagement with psychotherapy- dictated by physician);
12. Malignancies (basal cell carcinoma accepted);
13. Any contraindication for MRI.
14. New York Heart Association (NYHA) score of IV or hospitalisation from heart failure in the last 6 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population involves four groups: controls, OSA, COPD and overlap syndrome (OVS). All participants will meet all inclusion criteria for their group and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Scores on the Montreal Cognitive Assessment (MoCA) neuropsychological assessment for dementia risk. | Cross-sectional/baseline only
  MoCA scores of 18 to 25 indicate mild cognitive impairment, 10 to 17 indicate moderate cognitive impairment and scores below 10 indicate severe cognitive impairment.
  Associations between MoCA and night-time hypoxemia / sleep fragmentation in the entire sample.
Blood levels of amyloid beta (Aβ40/Aβ42 ratio). | Cross-sectional/baseline only
  Associations between blood levels of Aβ (Aβ40/Aβ42 ratio) and night-time hypoxemia / sleep fragmentation in the entire sample.

SECONDARY OUTCOMES:
Absolute Electroencephalographic (EEG) Power During Non-Rapid Eye Movement (NREM) Sleep. | Cross-sectional/baseline only
  Spectral power of delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges. Associations between absolute Electroencephalographic (EEG) Power During Non-Rapid Eye Movement (NREM) Sleep and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Brain tissue oxygenation during cognitive tasks and sleep. | Cross-sectional/baseline only
  Brain tissue oxygenation during sleep as measured by oxygenated and deoxygenated hemoglobin using functional Near Infrared Spectroscopy (fNIRS). Associations between brain tissue oxygenation and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Hypoxemia as measured by pulse oximetry. | Cross-sectional/baseline only
  Overnight hypoxemia measured by pulse oximetry through nocturnal readings of blood oxygen saturation (SpO2). Associations between night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Sleep Fragmentation | Cross-sectional/baseline only
  EEG arousal index (events per minute of total sleep time) measured during polysomnography. Associations between night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of premorbid functioning and preinjury through the Test of Premorbid Functioning (TOPF). | Cross-sectional/baseline only
  Neuropsychological Test: A z-score of -0.75 indicates low-average premorbid functioning, z= -1.40 indicates borderline poor premorbid functioning and inferior premorbid functioning spans from z=-2.05 to -3.65. Associations between TOPF scores and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of verbal learning and memory through the Rey Auditory Verbal Learning Test (RAVLT). | Cross-sectional/baseline only
  Neuropsychological Test: RAVLT scores between groups. Scores ≤ z= -1.0 across two domains indicate poor performance. Immediate verbal learning is assessed by summing trials 1 to 5, Learning is assessed from trial 5 minus trial 1, and Forgetting is assessed through trial five minus the delayed recall trial. Associations between RAVLT scores and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of mild forms of cognitive dysfunction through Delis Kaplan Executive Functioning System (D-CEFS) neuropsychological assessment. | Cross-sectional/baseline only
  Neuropsychological Test: Differences in scores between groups across the four trials. Greater time taken to complete the trials results in higher scores which indicate worse performance. Associations between D-CEFS scores night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of speed of processing and executive functioning through the Trail Making Test (TMT). | Cross-sectional/baseline only
  Neuropsychological Test: Differences in TMT scores between groups. Greater time taken to complete the tests results in higher scores which indicate worse performance. A TMT trial A score of ≥78 seconds and a TMT trial B score of ≥273 seconds indicates deficiency. Associations between TMT scores night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of verbal fluency through the Controlled Oral Word Association Test (COWAT). | Cross-sectional/baseline only
  Neuropsychological Test: Differences in the COWAT scores between groups. The more acceptable words stated across all four trials, the better the performance in the test. Associations between COWAT scores and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of attention, perceptual speed, motor speed and visual scanning through the Symbol Digits Modalities Test (SDMT). | Cross-sectional/baseline only
  Neuropsychological Test: Differences in the scores on the SDMT between groups. Scores on the SDMT range from 1 to 110, with higher scores indicating better performance over the 90-second trial. Associations between SDMT scores and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of fibrinogen. | Cross-sectional/baseline only
  Differences in the blood levels of fibrinogen between groups. Associations between fibrinogen and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of clusterin. | Cross-sectional/baseline only
  Differences in the blood levels of clusterin between groups. Associations between clusterin and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of 8-isoprostane | Cross-sectional/baseline only
  Differences in the blood levels of 8-isoprostane between groups. Associations between 8-isoprostane and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of C-reactive protein (CRP) | Cross-sectional/baseline only
  Differences in the blood levels of CRP between groups. Associations between CRP and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of erythrocyte sedimentation rate (ESR). | Cross-sectional/baseline only
  Differences in the blood levels of ESR between groups. Associations between ESR and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of plasma tau. | Cross-sectional/baseline only
  Differences in the blood levels of plasma tau between groups. Associations between plasma-tau and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of neurofilament light chain (NFL). | Cross-sectional/baseline only
  Differences in the blood levels of NFL between groups. Associations between NFL and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of Glial fibrillary acidic protein (GFAP). | Cross-sectional/baseline only
  Differences in the blood levels of GFAP between groups. Associations between GFAP and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of Apolipoprotein E gene (APOE-4). | Cross-sectional/baseline only
  Differences in the blood levels of APOE-4 between groups. Associations between APOE-4 and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of interleukin-8 (IL-8). | Cross-sectional/baseline only
  Differences in the blood levels of IL-8 between groups. Associations between IL-8 and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of interleukin-6 (IL-6). | Cross-sectional/baseline only
  Differences in the blood levels of IL-6 between groups. Associations between IL-6 and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of tumor necrosis factor alpha (TNFα). | Cross-sectional/baseline only
  Differences in the blood levels of TNFα between groups. Associations between TNFα and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Blood levels of amyloid beta (Aβ40/Aβ42 ratio). | Cross-sectional/baseline only
  Associations between blood levels of Aβ (Aβ40/Aβ42 ratio) and night-time hypoxemia / sleep fragmentation between groups.
Scores on the Montreal Cognitive Assessment (MoCA) neuropsychological assessment for dementia risk. | Cross-sectional/baseline only
  MoCA scores of 18 to 25 indicate mild cognitive impairment, 10 to 17 indicate moderate cognitive impairment and scores below 10 indicate severe cognitive impairment.
  Associations between MoCA and night-time hypoxemia / sleep fragmentation between groups.

OTHER OUTCOMES:
Brain structure: cortical thickness and volumetric brain maps | Cross-sectional/baseline only
  Brain MRI: T1-weighted imaging will be analysed to obtain individual cortical grey-matter thickness and volumetric maps. Associations of cortical thickness and brain-area volumes and night-time hypoxaemia / sleep fragmentation will be tested using permutation analysis of linear models on each vertex/voxel on the brain map, and corrected for multiple comparisons in the entire sample and between groups.
Brain structure: diffusion-weighted imaging | Cross-sectional/baseline only
  Brain MRI: Diffusion-weighted imaging will be analysed to obtain individual fractional anisotropy (FA) and mean diffusivity (MD) maps. Associations of FA and MD and night-time hypoxaemia / sleep fragmentation will be tested using permutation analysis of linear models on each voxel of the white-matter brain map, and corrected for multiple comparisons, in the entire sample and between groups.
Brain function: resting-state BOLD fMRI | Cross-sectional/baseline only
  Brain fMRI: Resting-state BOLD fMRI will be subjected to dual-regression independent component analysis to obtain individual spatial maps of multiple resting-state brain networks. The component weights of individual voxels will be associated with night-time hypoxaemia / sleep fragmentation using permutation analysis of linear models and corrected for multiple comparisons, in the entire sample and between groups.
Brain pathology: T1-weighted, T2-weighted, diffusion-weighted imaging, and FLAIR | Cross-sectional/baseline only
  Brain MRI: Structural scans will be used to identify potential brain pathology including, white-matter hyper- and hypo-intensities, lacunes, and potential infarcts or other potential ischaemic lesions. The number, type and anatomical location of these potential pathologies will be scored and associated with night-time hypoxaemia / sleep fragmentation using linear mixed models, in the entire sample and between groups.
Assessment of sensorimotor function and comprehension through the Motor Screening Task (MOT) of CANTAB. | Cross-sectional/baseline only
  CANTAB: Differences in scores on the MOT as measured by MOTML (the mean latency from display of a stimulus to the correct response). Greater scores indicate worse performance. Associations between MOT scores and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of processing and psychomotor speed through the Reaction Time (RTI) test of CANTAB. | Cross-sectional/baseline only
  CANTAB: Differences in scores on the RTI as measured by RTIFMDRT (the median time taken for the subject to select the target stimulus after releasing the button, calculated across all trials). Higher scores indicate worse performance. Associations between RTI scores night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of working memory and strategy through the Spatial Working Memory (SWM) test of CANTAB. | Cross-sectional/baseline only
  CANTAB: Differences in scores on the SWM as measured by SWMTE (total errors during the trials). Higher scores indicate worse performance. Associations between SWM scores and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Assessment of visual episodic memory through the Paired Associate Learning (PAL) test of CANTAB. | Cross-sectional/baseline only
  CANTAB: Differences in scores on the PAL as measured by PALTEA (The number of times the subject chose the incorrect box for a stimulus on assessment problems (PALTE), plus an adjustment for the estimated number of errors they would have made on any problems, attempts and recalls they did not reach). Higher scores indicate worse performance. Associations between PAL scores and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Sleep Spindles During Non-Rapid Eye Movement (NREM) Sleep | Cross-sectional/baseline only
  Sleep spindle and slow oscillation events in NREM sleep from in-laboratory overnight polysomnography. A sleep spindle and slow oscillation detection algorithm will be applied to electroencephalography (EEG) signals from polysomnography after artefacts are detected and removed. Associations between sleep spindles and slow oscillation events and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Traditional sleep staging. | Cross-sectional/baseline only
  Proportion of the sleep opportunity scored at the 5 stages (wake, and N1, N2, N3, and REM sleep) between lights out and lights on, and sleep onset, REM onset, sleep efficiency, measured using overnight in-laboratory polysomnography with high-density electroencephalogram (HdEEG), scored by a polysomnographic technician in accordance with American Academy of Sleep Medicine (AASM) Sleep Scoring criteria. Associations between traditional sleep staging and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Absolute Electroencephalography (EEG) Power During Rapid Eye Movement (REM) Sleep. | Cross-sectional/baseline only
  Spectral power of delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges. Power spectral analysis will be applied to EEG signals from polysomnography after artefacts are detected and removed. Associations between absolute Electroencephalography (EEG) Power During Rapid Eye Movement (REM) Sleep and night-time hypoxemia / sleep fragmentation in the entire sample and between groups.
Obstructive sleep apnoea (OSA) severity metrics | Cross-sectional/baseline only
  Apnoea-hypopnea index (AHI), oxygen desaturation index (ODI; 3%), oxygen saturation nadir, electroencephalogram (EEG) arousal index (number of arousals per hour of sleep). Associations between OSA severity metrics and night-time hypoxaemia/ sleep fragmentation in the entire sample and between groups.
Lung function as measured by clinical pulmonary function tests (PFT) | Cross-sectional/baseline only
  Pulmonary functioning as measured by traditional PFT (spirometry with pre and post bronchodilator, diffusing capacity of the lungs for carbon monoxide (DLCO), lung volumes and respiratory impedance (oscillometry) as dictated by the American Thoracic Society (ATS). Associations between lung function and night-time hypoxaemia/ sleep fragmentation in the entire sample and between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The Woolcock Institute of Medical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data pertaining to the OSA group will be shared with protocol number X22-0213 (Project: OSA-D; within The Woolcock Institute of Medical Research)
Time Frame: Data will become available upon collection. Data will be available for a minimum of 15 years.
Access Criteria: n=26 obstructive sleep apnoea (OSA) participants will meet all of the OSA inclusion criteria and none of the exclusion criteria.